CLINICAL TRIAL: NCT06979882
Title: Investigating Multigene Methylation Dynamics in Treatment Response Surveillance for Intestinal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20252140-F-1
Record Dates: First submitted 2025-04-23; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Intestinal Cancer
MeSH Terms: conditions — Intestinal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group one: Intestinal cancer patients undergoing primary surgical treatment
  Interventions: Other: Multi-gene methylation testing
- Group two: Intestinal cancer patients undergoing surgery following neoadjuvant therapy
  Interventions: Other: Multi-gene methylation testing
- Group three: Intestinal cancer patients undergoing active surveillance following neoadjuvant therapy
  Interventions: Other: Multi-gene methylation testing

INTERVENTIONS:
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group one
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group three
Other: Multi-gene methylation testing — Undergo multi-gene methylation testing in blood during follow-up
  Groups: Group two

SUMMARY:
The primary objective is to determine whether pretreatment-to-posttreatment changes in circulating multigene methylation levels correlate with objective response rates (ORR) assessed by contrast-enhanced CT/MRI and levels of serum tumor markers. Secondary endpoints include: (a) time-dependent association between methylation fluctuation patterns and progression-free survival (PFS), (b) comparative diagnostic accuracy of methylation indices versus conventional biomarkers, and (c) feasibility of using methylation thresholds to guide adaptive therapy modification.

ELIGIBILITY:
Inclusion Criteria:

Age at initial diagnosis: 18-75 years Histologically confirmed colorectal or small intestinal malignancy, with complete medical records, confirmed pathological diagnosis, and definitive staging data (TNM staging system) No history of other primary malignancies Absence of distant metastases (liver, lung, or other sites) confirmed by imaging examination (CT/MRI) No prior surgical resection, chemotherapy, or PD-1/PD-L1 immunotherapy before enrollment Availability of complete biospecimen information, including: Sample ID (medical record number), Demographic data (sex, age), Clinical diagnostic data, Tumor marker profiles (CEA, CA19-9, etc.)

Exclusion Criteria:

Life expectancy <6 months (as assessed by ECOG score ≥4 or Palliative Performance Scale ≤30%) Cognitive/psychiatric conditions: a. Legally incapacitated individuals without legal guardians, b. Active psychotic disorders (e.g., schizophrenia, bipolar disorder) or dementia (MMSE score <24) Investigator-determined exclusions

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 200
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2030-03-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Multi-gene methylation levels | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
Multi-gene methylation levels | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
Multi-gene methylation levels | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.

SECONDARY OUTCOMES:
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group one: Preoperative, 1 week, 1 month, 3 months, 6 months, 1 year, 1.5 years, 2 years, 3 years, 4 years, and 5 years postoperatively.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and postoperatively at 1 week, 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group two: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Tumor Markers (including CEA, AFP, CA125, CA19-9, CA72-4, etc.) results will be extracted from historical medical records, with test dates typically ranging from baseline (within 3 months pre-enrollment) to follow-up intervals aligned with standard clinical practice (e.g., every 3-6 months post-treatment). These time points may not synchronize with the methylation assessment schedule.
Imaging Examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Imaging examinations (including contrast-enhanced CT, PET/CT, ultrasound, X-ray, magnetic resonance imaging, etc.) results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.
Endoscope | Group three: pre-neoadjuvant therapy baseline, 1 week following neoadjuvant therapy, and post-neoadjuvant therapy at 1 month, 3 months, 6 months, 1 year, 18 months (1.5 years), 2 years, 3 years, 4 years, and 5 years.
  Endoscoping results will be collected from patient records. Imaging time points are determined by clinical needs (e.g., pre-treatment staging, 3-month post-treatment follow-up), with intervals independent of the methylation analysis schedule. The minimum interval between imaging and methylation sampling will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tangdu Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided